CLINICAL TRIAL: NCT02630368
Title: A Phase I/II Study of Metronomic Cyclophosphamide and Oncolytic Poxvirus JX-594 in Patients With Advanced Hormone-receptor Positive and Triple Negative Breast Cancer and Advanced Soft Tissue Sarcoma (METROmaJX)
Brief Title: A Study of Metronomic CP and JX-594 in Patients With Advanced Breast Cancer and Advanced Soft-tissue Sarcoma (METROmaJX)
Acronym: METROmaJX
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Bergonié (Other)
Collaborators: National Cancer Institute, France (Other Government); Fondation ARC (Other); Merck Sharp & Dohme LLC (Industry); Transgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IB 2014-02; 2014-001078-33 (EudraCT Number)
Record Dates: First submitted 2015-11-19; First posted 2015-12-15 (Estimated); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Solid Tumors; Soft-tissue Sarcoma; Breast Cancer
Keywords: Advanced Soft-tissue Sarcoma; Advanced Breast Cancer; Maximum Tolerated Dose; Efficacy and safety; Immunotherapy
MeSH Terms: conditions — Sarcoma; Breast Neoplasms | interventions — Cyclophosphamide; avelumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Experimental phase I dose escalating (Experimental): Prospective open-labeled phase I trial.
  Combination of cyclophosphamide and JX-594 dose escalation. Metronomic cyclophosphamide will be administered orally, 50 mg twice daily, one week on/one week off. JX-594 will be administered, as designated by assigned dose-level, intraveinously, on Days 8 and 22 of cycle 1, and on days 8 of each subsequent cycles. One cycle consits of 28 days.
  Number of subjects : 14
  Interventions: Drug: Cyclophosphamide and JX-594 dose escalation
- Experimental group soft-tissue sarcoma, treatment by JX-594 + Metronomic cyclophosphamide (Experimental): Randomized non comparative phase II clinical trial : Arm 1.
  Experimental phase II soft-tissue sarcoma :
  Combination of cyclophosphamide and JX-594. Metronomic cyclophosphamide will be administered orally, 50 mg twice daily, one week on/one week off. JX-594 will be administered, as the dose recommended in the experimental phase I dose escalating study, intraveinously, on Days 8 and 22 of cycle 1, and on days 8 of each subsequent cycles. One cycle consits of 28 days.
  Number of subjects : 48
  Interventions: Drug: Cyclophosphamide and JX-594
- Control group soft-tissue sarcoma, treatment by JX-594 + Metronomic cyclophosphamide (Experimental): Randomized non comparative phase II clinical trial : Arm 2.
  Control-arm phase II soft-tissue sarcoma :
  Patients will be treated by metronomic cyclophosphamide. Cyclophosphamide will be administered 50 mg twice daily orally, one week on/one week off. One cycle consits of 28 days.
  Number of subjects : 24
  Interventions: Drug: Cyclophosphamide
- Experimental group breast cancer, treatment by JX-594 + Metronomic cyclophosphamide (Experimental): Single-arm phase II clinical trial.
  Experimental phase II Group breast cancer :
  Combination of cyclophosphamide and JX-594. Metronomic cyclophosphamide will be administered orally, 50 mg twice daily, one week on/one week off. JX-594 will be administered, as the dose recommended in the experimental phase I dose escalating study, intraveinously, on Days 8 and 22 of cycle 1, and on days 8 of each subsequent cycles. One cycle consits of 28 days.
  Number of subjects : 32
  Interventions: Drug: Cyclophosphamide and JX-594
- Experimental group soft-tissue sarcoma, treatment by Avelumab + ITJX-594 + Metronomic CP (Experimental): Experimental phase II soft-tissue sarcoma :
  Combination of avelumab in combination with intratumoral JX-594 and metronomic cyclophosphamide.
  Avelumab will be administered by intravenous infusion every 2 weeks, starting at Day 15 of cycle 1.
  Cyclophosphamide wil be administered orally, 50 mg twice daily, one Week on/one Week off, starting 7 days prior to cycle 1 day 1 ("impregnation phase").
  JX-594 will be administered by intratumoral injection on day 1 of cycle 1, every 2 weeks, for a maximum of 4 injections.
  Number of subjects : 47
  Interventions: Drug: Avelumab and JX-594 and Cyclophosphamide
- Experimental group breast cancer, treatment by Avelumab + IT JX-594 + Metronomic CP (Experimental): Experimental phase II breast cancer :
  Combination of avelumab in combination with intratumoral JX-594 and metronomic cyclophosphamide.
  Avelumab will be administered by intravenous infusion every 2 weeks, starting at Day 15 of cycle 1.
  Cyclophosphamide wil be administered orally, 50 mg twice daily, one Week on/one Week off, starting 7 days prior to cycle 1 day 1 ("impregnation phase").
  JX-594 will be administered by intratumoral injection on day 1 of cycle 1, every 2 weeks, for a maximum of 4 injections.
  Number of subjects : 32
  Interventions: Drug: Avelumab and JX-594 and Cyclophosphamide

INTERVENTIONS:
Drug: Cyclophosphamide and JX-594 dose escalation — Metronomic cyclophosphamide will be administered orally, 50 mg twice daily, one week on/one week off. JX-594 will be administered, as designated by assigned dose-level, intraveinously, on Days 8 and 22 of cycle 1, and on days 8 of each subsequent cycles. One cycle consits of 28 days.
  Other Names: Brand name : ENDOXAN; Brand name: Pexa-Vec
  Arms: Experimental phase I dose escalating
Drug: Cyclophosphamide and JX-594 — Metronomic cyclophosphamide will be administered orally, 50 mg twice daily, one week on/one week off. JX-594 will be administered, as the dose recommended in the experimental phase I dose escalating study, intraveinously, on Days 8 and 22 of cycle 1, and on days 8 of each subsequent cycles. One cycle consits of 28 days.
  Other Names: Brand name : ENDOXAN; Brand name: Pexa-Vec
  Arms: Experimental group breast cancer, treatment by JX-594 + Metronomic cyclophosphamide; Experimental group soft-tissue sarcoma, treatment by JX-594 + Metronomic cyclophosphamide
Drug: Cyclophosphamide — Metronomic cyclophosphamide will be administered orally, 50 mg twice daily, one week on/one week off.
  Other Names: Brand name : ENDOXAN
  Arms: Control group soft-tissue sarcoma, treatment by JX-594 + Metronomic cyclophosphamide
Drug: Avelumab and JX-594 and Cyclophosphamide — Avelumab will be administered by intravenous infusion (10 mg/kg) every 2 weeks, starting at Day 15 of cycle 1.
  Cyclophosphamide wil be administered bi-daily (50 mg x 2), starting 7 days prior to cycle 1 day 1 ("impregnation phase") and given on a week on/week off schedule.
  JX-594 will be administered by intratumoral injection (1 x109 p.f.u) on day 1 of cycle 1, every 2 weeks, for a maximum of 4 injections .
  Other Names: Brand name: ENDOXAN; Brand name: Pexa-Vec; Brand name: Avelumab
  Arms: Experimental group breast cancer, treatment by Avelumab + IT JX-594 + Metronomic CP; Experimental group soft-tissue sarcoma, treatment by Avelumab + ITJX-594 + Metronomic CP

SUMMARY:
Assessment of the efficacy and safety of JX-594 and metronomic cyclophosphamide in patients with advanced soft-tissue sarcoma and advanced breast cancer, once the Maximum Tolerated Dose have been determined (phase I trial).

Phase I study: this is a prospective open-labeled phase I trial based on a dose escalating study design assessing two dose levels of JX594 when prescribed in combination with metronomic cyclophosphamide.

Phase II trials with two treatments strategies:

Metronomic CP + JX-594: phase II study sarcoma: this is a monocentric, randomized two-arm non comparative phase 2 study assessing efficacy and safety of JX-594 in association with metronomic cyclophosphamide in patients with advanced soft-tissue sarcoma.

Metronomic CP + JX-594: phase II study breast cancer: this is a monocentric, single-arm phase II study, assessing efficacy and safety of JX-594 in association with metronomic cyclophosphamide in patients with advanced breast cancer.

Metronomic CP + JX-594 + Avelumab: phase II study sarcoma: this is a monocentric, single arm phase II study assessing efficacy and safety of avelumab in combination with IT JX-594 and metronomic cyclophosphamide in patients with advanced soft-tissue sarcoma.

Metronomic CP + JX-594 + Avelumab:: phase II study breast cancer: this is a monocentric, single-arm phase II study, assessing efficacy and safety of avelumab in combination with IT JX-594 and metronomic cyclophosphamide in patients with advanced breast cancer.

DETAILED DESCRIPTION:
For the phase I study, this is a prospective open-label phase I trial based on a dose escalating study design assessing two dose level of JX-594 when associated to metronomic cyclophosphamide.

For the phase II study, two distincts treatment strategies will be evaluated.

First, treatment by JX-594 and metronomic cyclophosphamide:

* stratum soft-tissue sarcoma, this is a monocenter, randomized non comparative phase II clinical trial. This phase II trial was based on an optimal 2-stage Simon's design. Randomization 2:1 with 2 patients randomized in experimental arm n°1 (association of metronomic cyclophosphamide and JX-594) and 1 patient randomized in control arm n°2 (treatment by metronomic cyclophosphamide alone).
* stratum breast cancer, this is a monocenter, one-arm phase II clinical trial, based on two-stage optimal Simon's design (association of metronomic cyclophosphamide and JX-594).

Second, treatment by Avelumab, intratumoral JX-594 and metronomic cyclophosphamide:

* stratum soft-tissue sarcoma, this is a monocenter, single arm phase II clinical trial based on an optimal 2-stage Simon's design.
* stratum breast cancer, this is a monocenter, one-arm phase II clinical trial, based on two-stage optimal Simon's design).

ELIGIBILITY:
Main Inclusion Criteria:

1. Histology:

   * Phase Ib : Patient with histologically confirmed solid tumor
   * Phase II :

     * Patients with histologically confirmed HER2 negative breast cancer (treatment by CP+JX-594), or triple negative (treatment by avelumab + CP+JX-594)
     * Patients with histologically confirmed soft tissue sarcoma confirmed by the RRePS Network, b)Progressive disease or relapse, after standard therapy according to RECIST v1.1 criteria diagnosed on the basis of two CT scan or MRI obtained at an interval less than 6 months in the period of 12 months prior to inclusion and confirmed by central review
2. Metastatic or unresectable locally advanced disease
3. Age ≥ 18 years
4. ECOG ≤ 1 (Phase Ib), ≤ 2 (Phase II JX+CP) and ≤ 1 (Phase II avelumab+JX+CP).
5. Life expectancy > 3 months,
6. Measurable disease according to RECIST v1.1 outside any previously irradiated field. For patients treated by avelumab+JX+CP, at least one injectable site ≥ 2 cm and ≤ 8 cm in diameter and one distant non-injected measurable site (target site)
7. At least three weeks since last chemotherapy, immunotherapy or any other pharmacological treatment and/or radiotherapy.
8. Adequate hematological, renal, metabolic and hepatic functions.
9. Women of childbearing potential must have a negative serum pregnancy test before study entry. Both women and men must agree to use a medically acceptable method of contraception throughout the treatment period and for six months after discontinuation of treatment.
10. Patients informed of risks regarding drug interactions: patients receiving any substances that are inhibitors or inducers of CYP450 2B6 are ineligible
11. Voluntarily signed and dated written informed consent prior to any study specific procedure.
12. Patients with a social security in compliance with the French law.

Main Exclusion Criteria:

1. Previous treatment with JX-594 or other vaccina vector based treatment .
2. Concomitant diseases/conditions (non exhaustive list):

   1. Clinically significant immunodeficiency, such as HIV or active Hepatite B or C
   2. Any other major illness that, in the Investigator's judgment, will substantially increase the risk associated with the patient's participation in this study.
   3. History of severe exfoliative skins condition requiring systemic treatment for more than 4 weeks in the last two years.
   4. active autoimmune disease for patients treated by avelumab
3. Active central nervous system metastasis (CNS)
4. Participation to a study involving a medical or therapeutic intervention in the last 30 days.
5. Previous enrolment in the present study.
6. Patient unable to follow and comply with the study procedures because of any geographical, social or psychological reasons.
7. Known hypersensitivity to any involved study drug or any of its formulation components.
8. Use of steroids (any route of administration), interferon/pegylated interferon or ribavirin that cannot be discontinued within 14 days prior to any JX-594 dose.
9. No prior malignancy except for the following: adequately treated basal or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage 1 or Stage 2 cancer from which the patient is currently in complete remission or any other cancer from which the patient has been disease-free for 3 years.
10. Active cardiovascular disease, including but not limited to significant coronary artery disease (e.g. requiring angioplasty or stenting) or congestive heart failure within the preceding 12 months. (treatment by CP+JX)
11. Inability to suspend treatment with anti-hypertensive medication for 48 hours prior to and 48 hours after all JX-594 treatments.
12. Pulse oximetry O2 saturation < 90% at rest on room air.
13. Experienced a severe systemic reaction or side-effect as result of previous smallpox vaccination.
14. Cardiac disease: LVEF out of normal limits ; cumulative dose of anthracyclines in excess of 450 mg/m²
15. Known urinary tract obstruction
16. Household contact exclusions for patients enrolled: children< 1 year old ; People with skin disease (e.g., eczema, atopic dermatitis and related diseases…), Immunocompromised hosts (severe deficiencies in cell-mediated immunity, including AIDS, organ transplant recipients, hematologic malignancies)
17. Vaccination within 4 weeks of the first dose of study treatment and while on trial is prohibited except for administration of inactivated vaccines.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Estimated)
Dates: Start 2015-09-18 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Phase Ib : Maximum Tolerated Dose evaluated on the first cycle (D1 to D28) of the combination of JX-594 And metronomic cyclophosphamide | during the first cycle (28 days)
  the MTD is defined as the highest dose at which no more than 1 in 6 of the patients in the cohort experienced a DLT in the first treatment cycle
Phase II : Advanced soft-tissue sarcoma: Assessment of the antitumor activity of the association of JX-594 and metronomic cyclophosphamide based on 6 month non-progression (CR, PR or SD more than 24 weeks) following RECIST v1.1 criteria | Phase II : 6 months after the beginning of treatment
  Non-progression is defined as complete or partial response or stable disease, as per RECIST v1.1
Phase II : Advanced Breast cancer: Assessment of the antitumor activity of the association of JX-594 and metronomic cyclophosphamide Efficacy will be defined based on objective response under treatment (CR or PR) following RECIST v1.1 criteria | Phase II : 6 months after the beginning of treatment
  Objective response is defined as complete or partial response as per RECIST v1.1
Phase II : Advanced soft-tissue sarcoma: Assessment of the antitumor activity of Avelumab in combination with IT JX-594 and metronomic cyclophosphamide based on 6 month non-progression (CR, PR or SD more than 24 weeks) following RECIST v1.1 criteria | Phase II : 6 months after the beginning of treatment
  Non-progression is defined as complete or partial response or stable disease, as per RECIST v1.1
Phase II : Advanced Breast cancer: Assessment of the antitumor activity of avelumab in combination with IT JX-594 and metronomic cyclophosphamide Efficacy will be defined based on objective response under treatment following RECIST v1.1 criteria | Phase II : 6 months after the beginning of treatment
  Objective response is defined as complete or partial response as per RECIST v1.1

SECONDARY OUTCOMES:
Phase Ib : Recommended Phase II dose (RP2D) of the association of JX-594 and metronomic cyclophosphamide | Phase Ib : Throughout the 6 months of treatment period
  Data from all cycles will be used to define the dose level of JX-594 to be recommended for further investigations in phase II
Phase Ib: Objective response under treatment as per RECIST V1.1 | an average of 6 months
  Objective response is defined as complete or partial response as per RECIST v1.1
Phase Ib: Best overall response as per RECIST V1.1 | an average of 6 months
  - Best overall response is defined as the best response recorded from the start of the study treatment until the end of treatment taking into account any requirement for confirmation (as per RECIST v1.1).
Phase Ib: 6-months non-progression as per RECIST V1.1 | 6-months after the beginning of treatment
  Non-progression is defined as complete or partial response or stable disease, as per RECIST v1.1
Phase Ib: 1-year progression-free survival as per RECIST V1.1 | 1-year after the beginning of treatment
  PFS defined as the time from study treatment initiation to the first occurrence of disease progression or death (of any cause)
Phase Ib: 2-year progression-free survival as per RECIST V1.1 | 2-year after the beginning of treatment
  PFS defined as the time from study treatment initiation to the first occurrence of disease progression or death (of any cause)
Phase Ib : Pharmacokinetics (PK): PK measurements expressed as Area Under the curve forJX-594 | Day 8 of cycle 1, Day 15 of cycle 1, Day 22 of cycle 1, Day 1 of cycle 2, Day 8 of cycle 2, Day 22 of cycle 2, Day 8 of cycle 3, Day 8 of cycle 4, Day 8 of cycle 6 (Each cycle = 28 days)
Phase Ib : Pharmacokinetics (PK): PK measurements expressed as half-life forJX-594 | Day 8 of cycle 1, Day 15 of cycle 1, Day 22 of cycle 1, Day 1 of cycle 2, Day 8 of cycle 2, Day 22 of cycle 2, Day 8 of cycle 3, Day 8 of cycle 4, Day 8 of cycle 6 (Each cycle = 28 days)
Phase Ib : Pharmacokinetics (PK): PK measurements expressed as Concentration peak forJX-594 | Day 8 of cycle 1, Day 15 of cycle 1, Day 22 of cycle 1, Day 1 of cycle 2, Day 8 of cycle 2, Day 22 of cycle 2, Day 8 of cycle 3, Day 8 of cycle 4, Day 8 of cycle 6 (Each cycle = 28 days)
Phase Ib : Dose-Limiting toxicity of the association of JX-594 and metronomic cyclophosphamide | during the first cycle (cycle = 28 days)
Phase Ib : Predictive biomarkers analysis (cytokines levels) | baseline, day 8 of cycle 1, day 22 of cycle 1, day 8 of cycle 2, day 8 of cycle 4, day 8 of cycle 6. Each cycle = 28 days
Phase Ib : Predictive biomarkers analysis (lymphocytes levels) | baseline, day 8 of cycle 1, day 22 of cycle 1, day 8 of cycle 2, day 8 of cycle 4, day 8 of cycle 6. Each cycle = 28 days
Phase II : Best overall response defined as per RECIST v1.1 criteria | an average of 6 months
  Best overall response is defined as the best response recorded from the start of the study treatment until the end of treatment taking into account any requirement for confirmation (as per RECIST v1.1).
Phase II : For sarcoma only: objective response following CHOI criteria | an average of 6 months
Phase II : For sarcoma only: best overall response following CHOI criteria | an average of 6 months
Phase II : For sarcoma only: 6- month non-progression following CHOI criteria | 6-months after the beginning of treatment
Phase II : 1-year Progression-Free Survival (PFS) defined as the time from study treatment initiation to the first occurrence of disease progression or death (of any cause), whichever occurs first | one year after the beginning of treatment
  PFS defined as the time from study treatment initiation to the first occurrence of disease progression or death (of any cause)
Phase II : 2-year Progression-Free Survival (PFS) defined as the time from study treatment initiation to the first occurrence of disease progression or death (of any cause), whichever occurs first | two years the beginning of treatment
  PFS defined as the time from study treatment initiation to the first occurrence of disease progression or death (of any cause)
Phase II : 1-year Overall Survial (OS) defined as the time from study treatment initiation to death (of any cause) | one year after the beginning of treatment
  OS defined as the time from study treatment initiation to death (of any cause)
Phase II : 2-year Overall Survial (OS) defined as the time from study treatment initiation to death (of any cause) | two year after the beginning of treatment
  OS defined as the time from study treatment initiation to death (of any cause)
Phase II : Toxicity graded using the common toxicity criteria from the NCI v4.0 | an average of 6 months
  assessef with NCI-CTCAE V4
Predictive biomarkers (cytokines level) | baseline, day 8 of cycle 1, day 22 of cycle 1, day 8 of cycle 2, day 8 of cycle 4, day 8 of cycle 6. Each cycle = 28 days
Predictive biomarkers (lymphocytes level) | baseline, day 8 of cycle 1, day 22 of cycle 1, day 8 of cycle 2, day 8 of cycle 4, day 8 of cycle 6. Each cycle = 28 days
Phase II : Relationship between levels of anti-JX-594 antibodies and efficacy of CP + JX-594 in terms of 6-month non progression for sarcoma (as per RECIST V1.1) | Six months after the beginning of treatment
Phase II : Relationship between levels of anti-JX-594 antibodies and efficacy of CP + JX-594 in terms of objective response for breast cancer (as per RECIST V1.1) | an average of 6 months
Phase II : Relationship between activation of the pRB/E2F/TK pathway and efficacy of CP + JX-594 on available archived tumor tissue in terms of 6- month non progression for sarcoma (as per RECIST V1.1) | Phase II : Six months after the beginning of treatment
Phase II : Relationship between activation of the pRB/E2F/TK pathway and efficacy of CP + JX-594 on available archived tumor tissue in terms objective response for breast cancer (as per RECIST V1.1) | an average of 6 months
Phase II Soft-tissue sarcoma: antitumor actiivty of avelumab in combination with IT JX-594 and metronomic CP in terms of best overall response | an average of 6 months
  - Best overall response is defined as the best response recorded from the start of the study treatment until the end of treatment taking into account any requirement for confirmation (as per RECIST v1.1)
Phase II Breast cancer: antitumor actiivty of avelumab in combination with IT JX-594 and metronomic CP in terms of best overall response | an average of 6 months
  - Best overall response is defined as the best response recorded from the start of the study treatment until the end of treatment taking into account any requirement for confirmation (as per RECIST v1.1)
Phase II Breast cancer: antitumor actiivty of avelumab in combination with IT JX-594 and metronomic CP in terms of 6-month non-progression | 6 months
  Non-progression is defined as complete or partial response or stable disease, as per RECIST v1.1
Phase II Soft-tissue sarcoma: antitumor actiivty of avelumab in combination with IT JX-594 and metronomic CP in terms of objective response Under treatment | an average of 6 months
  Objective response is defined as complete or partial response as per RECIST v1.1
Phase II Soft-tissue sarcoma: antitumor actiivty of avelumab in combination with IT JX-594 and metronomic CP in terms of 1-year progression-free survival | 1 year
  PFS defined as the time from study treatment initiation to the first occurrence of disease progression or death (of any cause)
Phase II Breast cancer: antitumor actiivty of avelumab in combination with IT JX-594 and metronomic CP in terms of 1-year progression-free survival | 1 year
  PFS defined as the time from study treatment initiation to the first occurrence of disease progression or death (of any cause)
Phase II Soft-tissue sarcoma: antitumor actiivty of avelumab in combination with IT JX-594 and metronomic CP in terms of 2-year progression-free survival | 2 years
  PFS defined as the time from study treatment initiation to the first occurrence of disease progression or death (of any cause)
Phase II Breast cancer: antitumor activity of avelumab in combination with IT JX-594 and metronomic CP in terms of 2-year progression-free survival | 2 years
  PFS defined as the time from study treatment initiation to the first occurrence of disease progression or death (of any cause)
Phase II Soft-tissue sarcoma: antitumor activity of avelumab in combination with IT JX-594 and metronomic CP in terms of 1-year overall survival | 1 year
  OS defined as the time from study treatment initiation to death (of any cause)
Phase II Breast cancer: antitumor activity of avelumab in combination with IT JX-594 and metronomic CP in terms of 1-year overall survival | 1 year
  OS defined as the time from study treatment initiation to death (of any cause)
Phase II Soft-tissue sarcoma: antitumor activity of avelumab in combination with IT JX-594 and metronomic CP in terms of 2-year overall survival | 2 year
  OS defined as the time from study treatment initiation to death (of any cause)
Phase II Breast cancer: antitumor activity of avelumab in combination with IT JX-594 and metronomic CP in terms of 2-year overall survival | 2 year
  OS defined as the time from study treatment initiation to death (of any cause)
Phase II Soft-tissue sarcoma: safety profile of avelumab in combination with IT JX-594 and metronomic CP | throughout the treatment period, an expected average of 6 months
  Safety profile will be assessed as per NCI-CTCAE v5
Phase II breast cancer: safety profile of avelumab in combination with IT JX-594 and metronomic CP | throughout the treatment period, an expected average of 6 months
  Safety profile will be assessed as per NCI-CTCAE v5

CONTACTS AND LOCATIONS:
Overall Officials: Antoine ITALIANO, MD, PhD, Study Chair — Institut Bergonié
Locations (1):
- Institut Bergonie, Bordeaux, France